CLINICAL TRIAL: NCT04431440
Title: Bactericidal Effect of Silver Nanoparticles on Methecillin and Vancomycin Resistant Staphylococcus. Aureus (MRSA) Isolated From Critically Ill Patients
Brief Title: Silver Nanoparticles in Multidrug Resistant Bacteria
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia, Assiut University
Other Study IDs: XXXXX
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Multidrug Resistent Bacteria
MeSH Terms: interventions — colloidal silver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methicillin resistant staphylococcus aureus
  Interventions: Other: silver nanoparticles
- vancomycin resistent staphylococcus aureus
  Interventions: Other: silver nanoparticles

INTERVENTIONS:
Other: silver nanoparticles — effect silver nanoparticles will be examined on multidrug resistant bacteria

SUMMARY:
Recently, silver nanoparticles (AgNPs) have been widely used in various applications as antimicrobial agents, anticancer, diagnostics, biomarkers, cell labels, and drug delivery systems for the treatment of various diseases. The present study investigated the bactericidal effect of AgNPs against Methecillin Resistant Staph. aureus (MRSA) and Vancomycin resistant Staph aureus (VRSA)

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patients

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: critically ill patients
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
bactericidal effect of silver nanoparticles on multidrug resistant bacteria | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elsawy S, Elsherif WM, Hamed R. Effect of silver nanoparticles on vancomycin resistant Staphylococcus aureus infection in critically ill patients. Pathog Glob Health. 2021 Jul;115(5):315-324. doi: 10.1080/20477724.2021.1914412. Epub 2021 Apr 19. PMID 33872131